CLINICAL TRIAL: NCT05545917
Title: Advanced Practice Physiotherapy Care in Emergency Departments for Patients With Musculoskeletal Disorders: A Pragmatic Cluster Randomized Controlled Trial and Cost Analysis
Brief Title: Advanced Practice Physiotherapy Care in Emergency Departments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Francois Desmeules, Full professor, Université de Montréal and Maisonneuve-Rosemont Hospital research center, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: RCT ED Canada
Record Dates: First submitted 2022-08-04; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Diseases or Conditions; Emergency Department; Physiotherapy
Keywords: Emergency department; Physiotherapist; Primary care; Musculoskeletal Disorders; Advanced practice physiotherapy
MeSH Terms: conditions — Musculoskeletal Diseases; Emergencies

STUDY DESIGN:
Intervention Model Description: Step wedge RCT
Who Masked: Investigator
Masking Description: Neither participants nor providers (PTs and physicians) will be blinded in this study in the context of this pragmatic RCT. An independent statistician not involved in any other parts of this trial and blinded to the participants' allocation, will conduct the statistical analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP care (Experimental): The experimental arm will receive advanced practice physiotherapy care.
  Interventions: Other: Experimental: APP care
- Usual physician care (Active Comparator): The control arm will receive usual ED physician care delivered only by an ED physician.
  Interventions: Other: Control - Usual physician care

INTERVENTIONS:
Other: Experimental: APP care — The experimental arm will receive advanced physiotherapy care (APP) care. Patients will be independently managed (assessment and intervention) by a PT. The PT will make a diagnosis and initiate an intervention plan (e.g. education and exercise). If relevant, the PT will make recommendations for medical imaging tests or medication. PTs will also recommend the proper discharge from the emergency department (ED), such as hospitalization, discharge without medical consultation/follow-up or discharge with a medical follow-up or rehabilitation in an outpatient setting.
  Arms: APP care
Other: Control - Usual physician care — The control arm will receive usual ED physician care delivered only by an ED physician. This will include independent assessment, treatment and discharge by an ED physician with no physiotherapy within the ED but physician's referral to outpatient physiotherapy or other professionals/medical specialists will be possible; overall care offered by the ED physician will not be standardized but will be systematically documented.
  Arms: Usual physician care

SUMMARY:
Overcrowding in emergency departments (ED) is a major concern worldwide. Recent reports show that Canada has among the longest ED waiting times and limited access to care has been associated with poorer outcomes for many patients. Patients suffering from musculoskeletal disorders (MSKD) represent at least 25% of all ED visits and this number is expected to increase with the aging population. New collaborative models of care have been emerging in various settings, such as EDs, and physiotherapists (PT) have been identified as expert clinicians to care for patients with MSKD. These advanced practice physiotherapy (APP) models of care often allow for a more extended scope of practice for PTs in which they have direct access to patients without a physician referral, triage patients and sometimes prescribe medical imaging or medication. ED APP has emerged as a promising new ED model of care, but evidence of the efficacy and safety of such models is still limited. Only a few RCTs have been conducted and no studies have assessed the efficacy or cost-utility of physiotherapy models of care for patients with MSKD in Canadian EDs. Evaluation of the benefits of such models is highly context-dependent and systematic evaluation of these models is warranted to support further implementation in Canada.

The aim of this multicenter stepped-wedge cluster RCT and cost analysis is to compare the effectiveness of a direct access APP model of care compared to usual physician ED care for persons presenting to an ED with a MSKD, in terms of pain, function, health care resources utilization and costs.

Evidence-based development of new APP models of care in EDs could help improve access and quality of care for Canadians, thus relieving some of the pressure on our healthcare system by providing new innovative pathways of access to care for these patients.

DETAILED DESCRIPTION:
Background: Overcrowding in emergency departments (ED) is a major concern and reports show that Canada has among the longest ED wait and length of stay times. Patients suffering from musculoskeletal disorders (MSKD) represent at least 25% of all ED visits and this number is expected to increase with the aging population. Physiotherapists (PT) have been identified as expert clinicians to care for patients with MSKD and new collaborative models of care involving PTs have been emerging in ED. Traditionally, PTs provide care in EDs only after physicians have assessed patients and made a referral for physiotherapy. More autonomous PT involvement in ED models of care allows for efficient collaborative practice with physicians and other professionals and can benefit ED performance, patient outcomes, as well as healthcare resource utilization. These advanced practice physiotherapy (APP) models of care often allow for a more extended scope of practice for PTs in which they have direct access to patients without a physician referral, triage patients and sometimes prescribe medical imaging or medication. ED APP has emerged as a promising new ED model of care, but evidence of the effectiveness of such models is limited. Only a few RCTs have been conducted and no studies have assessed the efficacy or cost-utility of APP models of care in Canadian EDs. Evaluation of the benefits of such models is highly context-dependent and systematic evaluation of these models is warranted to further support implementation in Canada. Objectives: To compare the effectiveness of a direct access APP model of care compared to usual physician ED care for persons presenting to an ED with a MSKD, in terms patient-related outcomes, health care resources utilization and costs.

Methods: This trial is a multicenter stepped-wedge cluster RCT with a cost analysis. Six EDs (clusters) will be randomized to a treatment sequence where patients will either be managed by an ED PT or receive usual ED physician care without the intervention of a PT. Seven hundred and forty four patients with a MSKD will be recruited. Main outcome measures will be the Brief Pain Inventory as well as the EQ-5D-5L for economic outcomes. Secondary measures will include validated self-reported disability questionnaires and other healthcare utilization outcomes such as prescription of imaging tests and medication. Adverse events and re-visits to ED will also be monitored. Outcomes will be collected at inclusion, at ED discharge and at 4, 12 and 26 weeks following the ED visit. Health care costs will be measured from the perspective of the public system using Time-Driven Activity Based Costing. Per-protocol and intention-to-treat analyses will be performed using linear mixed-models with a random effect for cluster and fixed effect for time. The diverse and complementary research team assembled has the required methodological expertise to successfully complete this trial and several knowledge users have been involved which assures the feasibility and maximizes the impacts of this project.

Discussion: MSKD not only represent a significant economic burden in Canada, but also have a significant impact on our health care system and the quality of life of Canadians. By providing an innovative pathway of access to care, APP care could help relieve pressure on Canadian ED and help provide efficient care for Canadians with MSKD.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with complaints related to common minor MSKD (e.g. back pain, joint sprain, osteoarthritis, muscle pain or tendinopathy) and being triaged by the triage nurse as level 3, 4, or 5 on the Canadian Triage and Acuity Scale (CTAS);
* aged 18 years or more;
* legally able to consent;
* able to understand/speak French or English;
* beneficiary of a provincial universal health insurance coverage.

Exclusion Criteria:

* having injury resulting from major trauma (e.g. high velocity trauma or major motor vehicle accident);
* presenting a major musculoskeletal injury (e.g. open fractures, unreduced dislocations, open wounds or a condition that needs an urgent surgical intervention);
* presenting red flags (e.g. progressive neurological deficits or infection-related symptoms);
* consulting for a diagnosed inflammatory arthritis or other active/unstable non-musculoskeletal condition (e.g. pulmonary, cardiac, digestive or psychiatric condition) and
* consulting for a work-related MSKD eligible for workers' compensation benefits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short form, Pain interference scale (BPI) | At inclusion and respectively at 4-, 12- and 26- weeks after inclusion
  The BPI is a self-administered questionnaire that includes seven items where the patient is asked to rate the impact of pain on various functional activities (pain interference scale) using a 10-point scale. The BPI is valid, reliable and responsive to change in MSKD populations. Change between different time points will be assessed.
Costs analyses | At inclusion
  For cost analyses, Time-Driven Activity Based Costing analyses to be used are based on combining process-mapping and resource level costing. The overarching objective is to calculate the costs of all resources consumed as a patient moves along a care pathway, which is determined via a collaboration between clinical and administrative staff and each step of the pathway represents direct and indirect resources consumed when providing patient care. The cost of all resources (personnel including salaries of PT and physicians, consumables, overhead, etc.) is calculated on a per minute basis (Capacity Cost Rate -CCR). The total cost of an episode of care is determined based on the type of resources utilized by a patient and the amount of time consumed. In addition to calculating costs per patient, this methodology will be applied at the 6 different sites and hence allowing us to map the care pathway used in all the different sites.
Costs analyses | At 4 weeks after inclusion
  For cost analyses, Time-Driven Activity Based Costing analyses to be used are based on combining process-mapping and resource level costing. The overarching objective is to calculate the costs of all resources consumed as a patient moves along a care pathway, which is determined via a collaboration between clinical and administrative staff and each step of the pathway represents direct and indirect resources consumed when providing patient care. The cost of all resources (personnel including salaries of PT and physicians, consumables, overhead, etc.) is calculated on a per minute basis (Capacity Cost Rate -CCR). The total cost of an episode of care is determined based on the type of resources utilized by a patient and the amount of time consumed. In addition to calculating costs per patient, this methodology will be applied at the 6 different sites and hence allowing us to map the care pathway used in all the different sites.
Costs analyses | At 12 weeks after inclusion
  For cost analyses, Time-Driven Activity Based Costing analyses to be used are based on combining process-mapping and resource level costing. The overarching objective is to calculate the costs of all resources consumed as a patient moves along a care pathway, which is determined via a collaboration between clinical and administrative staff and each step of the pathway represents direct and indirect resources consumed when providing patient care. The cost of all resources (personnel including salaries of PT and physicians, consumables, overhead, etc.) is calculated on a per minute basis (Capacity Cost Rate -CCR). The total cost of an episode of care is determined based on the type of resources utilized by a patient and the amount of time consumed. In addition to calculating costs per patient, this methodology will be applied at the 6 different sites and hence allowing us to map the care pathway used in all the different sites.
Costs analyses | At 26 weeks after inclusion
  For cost analyses, Time-Driven Activity Based Costing analyses to be used are based on combining process-mapping and resource level costing. The overarching objective is to calculate the costs of all resources consumed as a patient moves along a care pathway, which is determined via a collaboration between clinical and administrative staff and each step of the pathway represents direct and indirect resources consumed when providing patient care. The cost of all resources (personnel including salaries of PT and physicians, consumables, overhead, etc.) is calculated on a per minute basis (Capacity Cost Rate -CCR). The total cost of an episode of care is determined based on the type of resources utilized by a patient and the amount of time consumed. In addition to calculating costs per patient, this methodology will be applied at the 6 different sites and hence allowing us to map the care pathway used in all the different sites.

SECONDARY OUTCOMES:
Pain intensity | Following initial assessment by provider in the emergency department
  0-10 numerical pain scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain)
Disability questionnaires - Neck Disability Index (NDI) | At inclusion and respectively at 4-, 12- and 26- weeks after inclusion
  For participants presenting with neck disorders, the Neck Disability Index (NDI) questionnaire will be completed. The score ranges from 0 to 50, with higher scores associated with higher disability levels.
Disability questionnaires - Oswestry Disability Index (ODI) for back related disorders | At inclusion and respectively at 4-, 12- and 26- weeks after inclusion
  For participants presenting with back related disorders, the Oswestry Disability Index (ODI) will be completed. The total score ranges from 0% to 100%, with higher scores relating to higher disability levels.
Disability questionnaires - short version of the Disability of the Arm, Shoulder and Hand (Quick DASH) | At inclusion and respectively at 4-, 12- and 26- weeks after inclusion
  For participants presenting with upper limb disorders, the short version of the Disability of the Arm, Shoulder and Hand (Quick DASH) will be completed. The score ranges from 0 to 100, where a higher score indicates a greater level of disability.
Disability questionnaires - Lower Extremity Functional Scale (LEFS) | At inclusion and respectively at 4-, 12- and 26- weeks after inclusion
  For participants presenting with lower limb disorders, the Lower Extremity Functional Scale (LEFS) questionnaire will be completed. The score ranges from 0 to 80, with lower scores indicating lower function levels.
Patient satisfaction assessed by the visit-specific satisfaction questionnaire (VSQ-9) | Following initial assessment by provider in the emergency department
  To assess satisfaction with care, patients will be asked to complete a modified validated version of the 9-item visit-specific satisfaction questionnaire (VSQ-9). Scores can range for 7 to 35 and lower scores are associated with higher satisfaction rates.
Wait to initial assessment | At inclusion
  Chronometer / clock
Emergency department length of stay | At inclusion
  Chronometer / clock
Health care resource utilization outcomes | At 4-, 12- and 26- weeks after inclusion
  Treatment diary:
  Participants will be asked to complete a treatment diary regarding compliance with ED treatments and any health services or interventions they sought for their initial problem during the follow-up period
Health care resource utilization outcomes | Immediately after initial assessment by provider in the emergency department
  Standardized evaluation form:
  Providers will complete a standardized form following their assessment and interventions, indicating diagnoses, requests for additional medical imaging or laboratory tests (if relevant), treatment plan (e.g. conservative treatment options, medication or physiotherapy care), discharge plan and referral to other professional or medical specialists, if relevant.

CONTACTS AND LOCATIONS:
Overall Officials: François Desmeules, Principal Investigator — Maisonneuve-Rosemont Research Center; Kadija Perreault, Principal Investigator — Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale; Marcel Emond, Principal Investigator — CHU de Québec - Université Laval (CHUQ-UL)

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this trial will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After all analyses have been conducted and results published
Access Criteria: The data that support the findings of this trial will be available upon reasonable request.

REFERENCES:
- [Derived] Matifat E, Berger Pelletier E, Brison R, Hebert LJ, Roy JS, Woodhouse L, Berthelot S, Daoust R, Sirois MJ, Booth R, Gagnon R, Miller J, Tousignant-Laflamme Y, Emond M, Perreault K, Desmeules F. Advanced practice physiotherapy care in emergency departments for patients with musculoskeletal disorders: a pragmatic cluster randomized controlled trial and cost analysis. Trials. 2023 Feb 6;24(1):84. doi: 10.1186/s13063-023-07100-x. PMID 36747305